CLINICAL TRIAL: NCT04981509
Title: A Phase 2 Study of Bevacizumab, Erlotinib and Atezolizumab in Subjects With Advanced Hereditary Leiomyomatosis and Renal Cell Cancer (HLRCC) Associated or Sporadic Papillary Renal Cell Cancer
Brief Title: Testing of Bevacizumab, Erlotinib, and Atezolizumab in Combination for Advanced-Stage Kidney Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-07744; NCI-2021-07744 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10466 (Other: National Cancer Institute LAO); 10466 (Other: CTEP)
Record Dates: First submitted 2021-07-28; First posted 2021-07-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Hereditary Leiomyomatosis and Renal Cell Carcinoma; Papillary Renal Cell Carcinoma; Renal Cell Carcinoma; Sporadic Papillary Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Hereditary leiomyomatosis and renal cell cancer; Carcinoma, Renal Cell; Papillary renal cell carcinoma, sporadic | interventions — atezolizumab; Bevacizumab; Immunoglobulin G; Disulfides; Biopsy; Specimen Handling; Contrast Media; Erlotinib Hydrochloride; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (bevacizumab, atezolizumab, erlotinib) (Experimental): Patients receive bevacizumab IV over 30-90 minutes and atezolizumab IV over 30-60 minutes on day 1 of each cycle. Patients also receive erlotinib PO QD on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT with or without contrast and MRI throughout the trial. Patients undergo collection of blood throughout the trial, and may undergo a biopsy during screening, as well as a brain MRI/CT scan with contrast, bone scan, and/or F-18 sodium fluoride PET scan as clinically indicated.
  Interventions: Biological: Atezolizumab; Biological: Bevacizumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Computed Tomography with Contrast; Drug: Erlotinib; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Sodium Fluoride F-18

INTERVENTIONS:
Biological: Atezolizumab — Given PO
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT without contrast
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Computed Tomography with Contrast — Undergo CT with contrast
  Other Names: Contrast Enhanced Computed Tomography; CONTRAST ENHANCED CT SCAN; Contrast-enhanced Computed Tomography; CT Scan With Contrast; CT with Contrast
Drug: Erlotinib — Given PO
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Sodium Fluoride F-18 — Given F-18 sodium fluoride
  Other Names: 18 F-NaF; F-18 NaF; Fluorine F 18 Sodium Fluoride; NaF F18; Sodium Fluoride F18

SUMMARY:
This phase II trial studies the effects of combination therapy with bevacizumab, erlotinib, and atezolizumab in treating patients with hereditary leiomyomatosis and kidney cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Bevacizumab is in a class of medications called antiangiogenic agents. They work by stopping the formation of blood vessels that bring oxygen and nutrients to tumors. This may slow the growth and spread of tumors. Erlotinib is in a class of medications called kinase inhibitors. It works by blocking the action of a protein called EGFR that signals cancer cells to multiply. This helps slow or stop the spread of cancer cells. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Combination therapy with bevacizumab, erlotinib, and atezolizumab may stabilize or shrink advanced hereditary leiomyomatosis and kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the complete response (CR) rate according to standard Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) in patients with 1) advanced renal cell cancer (RCC) associated with hereditary leiomyomatosis and renal cell cancer (HLRCC) and 2) advanced sporadic/non-HLRCC papillary renal cell cancer treated with a combination of bevacizumab, erlotinib, and atezolizumab.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of the combination of bevacizumab, erlotinib, and atezolizumab.

II. To determine the objective response rate (ORR) as complete response (CR) + partial response (PR).

III. To determine disease control rate (DCR) - confirmed response, or stable disease (SD) lasting for at least 6 months.

IV. To assess progression-free survival time (PFS) according to RECIST 1.1. V. To assess overall survival (OS). VI. To assess the duration of response. VII. To assess response to treatment using immune-modified Response Evaluation Criteria in Solid Tumors (iRECIST).

EXPLORATORY OBJECTIVES:

I. To evaluate immunologic modulation associated with the administered treatment regimen, including:

Ia. Peripheral immune subset analysis before and on treatment; Ib. Evaluation of relevant soluble factors before and on treatment. (e.g., cytokine profiles); Ic. Tumor tissue immune infiltration cells before and after treatment (immune microenvironment, CD8/CD4/CD3 cells, T-cell receptor clonality); Id. Evaluation of tissue PDL1/PD1 expression and their correlation with outcome.

II. To assess specific genomic alterations (including fumarate hydratase [FH], NRF2 pathway) and determine if there is a correlation with clinical outcomes.

OUTLINE:

Patients receive bevacizumab intravenously (IV) over 30-90 minutes and atezolizumab IV over 30-60 minutes on day 1 of each cycle. Patients also receive erlotinib orally (PO) once daily (QD) on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) with or without contrast and magnetic resonance imaging (MRI) throughout the trial. Patients undergo collection of blood throughout the trial, and may undergo a biopsy during screening, as well as a brain MRI/CT scan with contrast, bone scan, and/or F-18 sodium fluoride positron emission tomography (PET) scan as clinically indicated.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have:

  * A diagnosis of HLRCC with a histologic or cytologic confirmation of RCC consistent with this diagnosis (Cohort 1) OR
  * Cytologically or histologically confirmed sporadic/non-HLRCC papillary renal cell carcinoma (presence of papillary component) (Cohort 2)
* Patients must have advanced RCC with measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with CT scan, MRI, or calipers by clinical exam. To be considered pathologically enlarged and measurable, a lymph node must be >= 15 mm (>= 1.5 cm) in short axis
* Patients must have received no more than two prior regimens targeting the VEGF pathway and no prior bevacizumab therapy in the metastatic/advanced setting. No prior treatment with PD-1 or PD-L1 inhibitors in the metastatic/advanced setting. No prior therapy is required for eligibility
* Age >= 12 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (< 3 x upper limit of reference range in patients with known/suspected Gilbert's disease)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (or =< 5 x upper limit of reference range if considered to be related to liver or bone metastases by the principal investigator [PI])
* Alkaline phosphatase =< 2.5 x institutional ULN (or =< 5 x upper limit of reference range if considered to be related to liver or bone metastases by the PI)

  * Note: For pediatric patients (< 18 years of age), ULN for alkaline phosphatase will be defined as 390 IU/L for males and 320 IU/L for females
* Glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2

  * Note: For pediatric patients (< 18 years of age) the following creatinine thresholds will be utilized. Patients with a creatinine that exceeds this threshold will require further testing with a confirmation of GFR >= 40 as determined by either 24-hour urine collection or with radioisotope based nuclear medicine evaluation
  * Age: 12 to < 13 years; Maximum serum creatinine (mg/dL): 1.2 (male); 1.2 (female)
  * Age: 13 to < 16 years; Maximum serum creatinine (mg/dL): 1.5 (male); 1.4 (female)
  * Age: 16 to < 18 years; Maximum serum creatinine (mg/dL): 1.7 (male); 1.4 (female)

    * The threshold creatinine values in this table were derived from the Schwartz formula for estimating GFR, utilizing child length and stature data published by the Centers for Disease Control and Prevention (CDC)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with an undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression/recurrence for >= 3 months and the patient no longer requires more than a physiologic dose of steroids
* Patients with a prior or concurrent invasive malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with a known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* The effects of study drugs on the developing human fetus are unknown. For this reason, all women and men of childbearing potential must agree to use adequate contraception (including but not limited to abstinence, barrier methods, hormonal contraceptives [birth control pills, injections, or implants], intrauterine device [IUD], tubal ligation, vasectomy) prior to study entry and for 6 months after completion of study therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, and 6 months after completion of study drugs administration
* Subjects must provide archival tissue block or unstained tumor tissue or be willing to undergo biopsy to collect samples for retrospective central pathology review
* The ability of subject or parent/guardian to understand and the willingness to sign a written informed consent document or subjects with impaired decision making capacity (IDMC) if they are represented by a legally authorized representative (LAR)

Exclusion Criteria:

* Any prior systemic therapy to treat the patient's kidney cancer within 4 weeks or, if known, 5 half-lives of the prior agent (whichever is shorter) prior to cycle 1 day 1
* Other prior therapies for kidney cancer: Radiotherapy < 2 weeks prior to cycle 1, day 1
* Major surgical procedure < 28 days before cycle 1, day 1. Surgical procedure change (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to initiation of study treatment, or anticipation of need for major surgical procedure during the course of the study. Surgical wounds must be healed prior to starting therapy. However, the following therapies are allowed:

  * Hormone-replacement therapy or oral contraceptives
  * Herbal therapy > 1 week prior to cycle 1, day 1. All herbal therapy must be discontinued at least 1 week prior to cycle 1, day 1
  * Palliative radiotherapy for bone metastases > 2 weeks prior to cycle 1, day 1
* Patients who have not recovered from adverse events due to prior systemic anti-cancer therapy (i.e., have residual toxicities > grade 1 of the Common Terminology Criteria for Adverse Events [CTCAE] version [v]5, pre-treatment baseline or to a level permitted under other sections of inclusion/exclusion criteria) with the exception of alopecia or electrolyte abnormalities that can be corrected to =< grade 1 prior to treatment initiation
* Treatment with any other investigational agent within 4 weeks prior to cycle 1, day 1
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or interleukin [IL]-2) within 6 weeks prior to cycle 1, day 1
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to cycle 1, day 1

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea or for purposes of pre-medication prior to radiology studies) may be enrolled
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Hypercalcemia > grade 1 of the CTCAE v5 that is not corrected prior to treatment initiation
* Patients taking bisphosphonate therapy for symptomatic hypercalcemia. Use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed
* History of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * The disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
    * No acute exacerbations of the underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug-induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Patients with active tuberculosis (TB) are excluded
* Severe infections within 4 weeks prior to cycle 1, day 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1, day 1 or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of atezolizumab

  * NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines and are not allowed. Influenza vaccination should be given during influenza season only (approximately October to March)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Poorly controlled hypertension with at least 2 occasions of elevated blood pressure within a week before treatment initiation (Adults: resting systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg. Pediatric [< 18 years old]: Blood pressure [BP] >= the 95th percentile for age, height, and sex on at least two occasions separated by a 24-hour period despite optimal medical management). History of hypertensive crisis or hypertensive encephalopathy
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* History of anaphylactic or severe allergic reactions attributed to compounds of similar chemical or biologic composition to the study agents
* Patients with myocardial infarction, gastrointestinal (GI) perforation/fistula, intraabdominal abscess, or cerebrovascular accidents within 6 months before cycle 1, day 1
* Documented baseline proteinuria > 1000 mg/day on 24-hour urine collection. Only patients with 1+ or greater proteinuria on urinalysis (UA) and a spot urine protein:creatinine ratio of > 0.5 will undergo a 24-hour urine collection for quantitation of proteinuria
* Pregnant women are excluded from this study because study drugs may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with study drugs, breastfeeding should be discontinued if the mother is treated with study drugs
* Serious, non-healing wound or ulcer; bone fracture within 3 months prior to treatment initiation
* Concomitant therapy with potent inhibitors of CYP450 3A4 (e.g. ketoconazole, verapamil, etc.) or potent CYP3A4 inducers or with potent CYP450 1A2 inhibitors (fluoroquinolone antibiotics including ciprofloxacin, levofloxacin, and norfloxacin; ticlopidine, cimetidine, amiodarone, etc.) who cannot discontinue or change these medications prior to the start of study treatment
* Patients who use tobacco or nicotine products and cannot stop their use of these products for the duration of study treatment
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to cycle 1, day 1
* History of or active hemoptysis within 1 month prior to cycle 1 day 1
* History of grade >= 4 venous thromboembolism
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation)
* Current or recent (< 10 days prior to initiation of study treatment) use of aspirin (> 325 mg/day), or clopidogrel (> 75 mg/day)

  * Note: The use of full-dose oral or parenteral anticoagulants for therapeutic purpose is permitted as long as the International Normalized Ratio (INR) and/or a partial thromboplastin time (PTT) is within therapeutic limits (according to institution standards) within 7 days prior to initiation of study treatment and the patient has been on a stable dose of anticoagulants for >= 2 weeks prior to initiation of study treatment. Prophylactic use of anticoagulants is allowed. However, the use of direct oral anticoagulant therapies such as dabigatran (Pradaxa [registered trademark]) and rivaroxaban (Xarelto [registered trademark]) may be used per PI discretion

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 28 days after treatment
  To determine the safety and tolerability of the combination of bevacizumab, erlotinib, and atezolizumab, the fraction of patients with a dose-limiting toxicity will be reported, along with the maximum grade and type of toxicity for each type noted. Note: In addition to adverse events in the entire study population, pediatric toxicities will also be reported and analyzed separately.
Objective response rate | Up to 2 years from study enrollment
  Defined as complete response (CR) + partial response (PR), the fraction with a response (CR+PR) will be reported separately by cohort, along with a 95% confidence interval.
Disease control rate | Up to 2 years from study enrollment
  Will be reported for patients with confirmed response, or stable disease (SD) lasting for at least 6 months. Will be reported separately by cohort, along with a 95% confidence interval.
Progression-free survival time (PFS) | Time from study treatment initiation until disease progression or death, assessed up to 2 years from study enrollment
  Assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, PFS will be determined using the Kaplan-Meier method, and the curves presented along with a 95% confidence interval on the median PFS, separately by cohort.
Overall survival (OS) | From study treatment initiation until death from any cause, assessed up to 2 years from study enrollment
  The Kaplan-Meier method will be used and the curves presented along with a 95% confidence interval on the median OS, separately by cohort.
Duration of response (DOR) | Length of time without disease progression or recurrence, up to 2 years from study enrollment
  The Kaplan-Meier method will be used and the curves presented along with a 95% confidence interval on the median DOR, separately by cohort.
Response to treatment | Assessed up to 2 years from study enrollment
  Response to treatment using immune-modified Response Evaluation Criteria in Solid Tumors (iRECIST), the fraction with a response (CR+PR) according to iRECIST will be reported separately by cohort, along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Ramaprasad Srinivasan, Principal Investigator — National Cancer Institute LAO
Locations (13):
- United States (13):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm